CLINICAL TRIAL: NCT00702936
Title: Telmisartan vs Ramipril for Reduction of Inflammation and Recruitment of Endothelial Progenitor Cells After Acute Coronary Syndrome
Brief Title: Telmisartan Versus Ramipril After Acute Coronary Syndrome
Acronym: TERACS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Catholic University of the Sacred Heart, Catholic University of the Sacred Heart
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILG-1
Record Dates: First submitted 2008-06-19; First posted 2008-06-20 (Estimated); Last update posted 2008-06-20 (Estimated); Status verified 2008-06

CONDITIONS: Acute Coronary Syndrome; Myocardial Infarction; Coronary Disease
MeSH Terms: conditions — Acute Coronary Syndrome; Myocardial Infarction; Coronary Disease | interventions — Telmisartan; Ramipril

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- R (Active Comparator): Twenty-five patients assigned to ramipril 5 mg daily
  Interventions: Drug: RAMIPRIL
- T (Active Comparator): Twenty-five patients assigned to Telmisartan 80 mg daily
  Interventions: Drug: TELMISARTAN

INTERVENTIONS:
Drug: TELMISARTAN — 80 mg daily
  Arms: T
Drug: RAMIPRIL — 5 mg daily
  Arms: R

SUMMARY:
The purpose of this study is to compare the antinflammatory and endothelial progenitor cell (EPC) mobilizing effect of Ramipril and Telmisartan in patients presenting with acute coronary syndrome

ELIGIBILITY:
Inclusion Criteria:

* Biochemical evidence of myocardial infarction as indicated by elevation of cTnT,
* presence of ECG ischemic changes,
* angiographic evidence of a primary coronary event, such as plaque erosion and/or rupture, fissuring, or dissection at coronary angiography,
* successful coronary revascularization of at least one culprit coronary vessel.

Exclusion Criteria:

* Age>80 years, current ACE inhibitor or ARB treatment,
* ejection fraction <35%, infarction secondary to ischemia due to an imbalance of O2 supply and demand,
* ECG abnormalities that could affect the recognition of ST segment shift,
* recent or chronic infective or inflammatory diseases,
* malignancy, and myocardial infarction,
* surgery or trauma in the previous month.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2007-11; Primary Completion 2008-08 (Estimated); Study Completion 2008-11 (Estimated)

PRIMARY OUTCOMES:
High sensitivity C-Reactive Protein | 20 days after hospital discharge

SECONDARY OUTCOMES:
Endothelial Progenitor Cells | 20 days after hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Italo Porto, MD, PhD, Principal Investigator — Catholic University of the Sacred Heart; Luca Di Vito, MD, Principal Investigator — Catholic University of the Sacred Heart
Locations (1):
- Catholic University of the Sacred Heart, Rome, Italy

REFERENCES:
- [Background] Biasucci LM, Lombardi M, Piro M, Di Giannuario G, Liuzzo G, Crea F. Irbesartan significantly reduces C reactive protein concentrations after 1 month of treatment in unstable angina. Heart. 2005 May;91(5):670-1. doi: 10.1136/hrt.2004.036509. No abstract available. PMID 15831660
- [Result] Liakishev AA. [Telmisartan, ramipril, or both in patients at high risk for vascular events. Results of the ONTARGET trial]. Kardiologiia. 2008;48(5):72. No abstract available. Russian. PMID 18537808
- [Derived] Porto I, Di Vito L, De Maria GL, Dato I, Tritarelli A, Leone AM, Niccoli G, Capogrossi MC, Biasucci LM, Crea F. Comparison of the effects of ramipril versus telmisartan on high-sensitivity C-reactive protein and endothelial progenitor cells after acute coronary syndrome. Am J Cardiol. 2009 Jun 1;103(11):1500-5. doi: 10.1016/j.amjcard.2009.01.370. PMID 19463506